CLINICAL TRIAL: NCT01420822
Title: Special Drug Use Investigation for ALLERMIST (Long Term)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113406
Record Dates: First submitted 2011-06-02; First posted 2011-08-22 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis | interventions — Fluticasone

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects prescribed ALLERMIST: Subjects with allergic rhinitis prescribed ALLERMIST during study period
  Interventions: Drug: Fluticasone

INTERVENTIONS:
Drug: Fluticasone — Collection of safety data

SUMMARY:
This post-marketing surveillance study is to investigate possible problems or questions in safety and efficacy of ALLERMIST Nasal Spray for long-term use in Japanese subjects with allergic rhinitis under the conditions of actual practical use.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of allergic rhinitis
* Use ALLERMIST for the first time
* Expected to use ALLERMIST for long-term (1 year).

Exclusion Criteria:

* Subjects with infection which fluticasone is not effective
* Subjects with deep mycosis
* Subjects with hypersensitivity to fluticasone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target subjects shall be those who with allergic rhinitis for which the indication of ALLERMIST has been approved and who are using ALLERMIST for the first time and also who are expected to use ALLERMIST for long-term (1 year).
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The number of incidence of adverse events in Japanese subjects treated with ALLERMIST Nasal Spray for long-term use | One year
Efficacy evaluation based on the subjective/objective symptom progresses in the period from the start of Allermist treatment to the end of the observation period | One year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline